CLINICAL TRIAL: NCT06220656
Title: ThyRoid Active Monitoring and Intervention Longitudinal (TRAIL) Study: Feasibility and Pilot
Brief Title: TRAIL Study: Feasibility and Pilot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: American College of Radiology (Other); Dartmouth College (Other)
Responsible Party: Principal Investigator, Louise Davies, Staff Physician - Section of Otolaryngology Head & Neck Surgery, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY02002058; 23DAV058 (Other: Dartmouth Cancer Center)
Record Dates: First submitted 2023-12-22; First posted 2024-01-24 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Thyroid Nodule; Thyroid Neoplasms; Thyroid Cancer
MeSH Terms: conditions — Thyroid Nodule; Thyroid Neoplasms | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate biopsy (usual care) (Experimental): The aim of biopsy is to sample the thyroid nodule so that it can be tested for cancer. A biopsy is done with a small needle in an office. If the biopsy result shows the nodule is unlikely to be cancer, the next step is check-ups every 6 months to a year for two years followed by additional checkups that occur less frequently.
  If the biopsy result shows the nodule may be cancerous, usual treatment is surgery to remove part or all of the thyroid gland. Afterwards, regular check-ups and ultrasounds follow. Surgery may be outpatient or overnight stay. Recovery takes a couple weeks or more. Time in the hospital and recovering depends on the type of operation and any side-effects.
  Interventions: Procedure: Biopsy
- Active monitoring, proceeding to biopsy if needed (Experimental): The aim of Active Monitoring is to monitor the thyroid nodule closely. An ultrasound and a check-up with a clinician are done every six months for two years, then less often after that.
  If no changes in the nodule or new abnormal lymph nodes are seen, Active Monitoring continues and surgery and its side-effects are avoided. If changes in the nodule are seen on ultrasound, they are explained at the visit. The doctor may recommend that continued Active Monitoring or recommend a biopsy to investigate the changes. The biopsy result may suggest Active Monitoring can be continued, or may indicate surgery should be done, as described above.
  Interventions: Procedure: Active Monitoring

INTERVENTIONS:
Procedure: Biopsy — Local anesthetic is usually given and a small needle is used to take cells from the thyroid under ultrasound guidance through several 'passes' and placed into specialized media for pathology evaluation.
  Arms: Immediate biopsy (usual care)
Procedure: Active Monitoring — Ultrasound and a check-up at 6 months. Depending on ultrasound results, either biopsy and further care (as for the treatment arm called 'biopsy'), or continue with active monitoring.
  Arms: Active monitoring, proceeding to biopsy if needed

SUMMARY:
This is a pilot study to compare two ways of managing newly identified thyroid nodules that are likely to be cancerous based on ultrasound result and which under usual care would undergo immediate biopsy.

The main goals of this pilot study are 1) compare anxiety at 6 months in each treatment arm using the validated instrument Anxiety-CA, 2) measure thyroid quality of life in each treatment arm

Participants will be randomized to one of two groups:

1. immediate biopsy (usual care)
2. Active monitoring (serial ultrasound based monitoring and close clinical follow-up)

ELIGIBILITY:
Inclusion Criteria:

* Participants must be ≥18 years of age.
* Participants must be able and willing to provide informed consent or have a surrogate capable of providing same.
* Participants must be absent of symptoms referable to the nodule: dysphagia or nodule physically visible and/or bothersome to patient.
* Participants' thyroid nodule must have a TI-RADS rating of 4 or 5.
* Participants thyroid nodule must be ≤2 cm in largest diameter.
* Participants must be being considered for biopsy.
* Participants with a prior history of papillary thyroid cancer are eligible.

Exclusion Criteria:

Patients who fall into one of the following categories will NOT be eligible for this study:

* Adults who are unable to provide informed consent.
* Patients for whom biopsy is not a consideration.
* Patients with a prior history of thyroid cancer other than papillary thyroid cancer.
* Patients with a history of radiation to the neck.
* Patients who are athyroidal (thyroid gland has been removed or patient has only lingual thyroid tissue).
* Patients who have ultrasound evidence of one or more of the following:
* Airway invasion of the nodule.
* Nodule adjacency to/invading the recurrent nerve.
* Extra-thyroidal invasion by the nodule.
* Patients who have metastasis to cervical lymph nodes (confirmed by needle biopsy if ultrasound suspicious), distant metastases, if identified) testing not required, not usual care)
* Patients who have already had a biopsy of the nodule being considered for inclusion in the study.

TRAIL Pilot Integrated QRI: Inclusion/Exclusion Criteria

Inclusion Criteria for Study Patient Participants:

* Participants must meet the eligibility requirements above and will be or have been approached about enrolling in the pilot study.
* Participants must be willing to allow audio recorder presence and / or willing to be interviewed by the QRI team.

Exclusion Criteria for Study Patient Participants:

-Patients who are not willing to allow audio recorder presence and/or not willing to be interviewed by QRI team will be excluded from this study.

Inclusion Criteria for Study Staff Participants:

* Staff must be willing to audio record their communications with patients about enrolling in the study.
* Staff must be willing to participate in interviews with QRI team about their views of the study.

Exclusion Criteria for Study Staff Participants:

-Staff members who are not willing to participate in audio taping of recruitment discussions and/or interviews with QRI team about their views of the study will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Rate of Anxiety at 6 months | 6 months after randomization
  Rate of anxiety will be measured using Anxiety-CA instrument PROMIS-Anxiety Short form. Each question has five response options ranging in value from one to five. (1 = never experiencing a type of distressing emotion; 5 = always feeling that emotion). To find the total raw score for a short form with all questions answered, sum the values of the response to each question. For the adult PROMIS Anxiety 7a short form, a raw score of 10 converts to a T-score of 46.7 with a standard error (SE) of 2.6.

SECONDARY OUTCOMES:
Representativeness of enrolled participants compared to eligible participants | 6 months after randomization.
  Representativeness will be compared in terms of age in years (continuous), biological male or female (categorical), and race/ethnicity (categorical).
Study Procedure compliance | 6 months after randomization
  Rate of completion of patient reported outcomes and number of participants who withdraw from study or are lost to follow-up.
Clinical outcomes: needle biopsy cytology results (if done), | 6 months after randomization.
  A needle biopsy is a procedure to obtain samples of tissue or cells from thyroid nodule or lymph nodes to reveal whether a nodule is a benign tumor or cancer. Bethesda classification (ordinal) will be used. The Bethesda system identifies six diagnostic categories on thyroid nodule cytopathology. Each category is linked to a malignancy risk. Categories are as follows: Category I (Nondiagnostic), Category II (Benign), Category III (Atypical of undetermined significance), Category IV (Suspicious for follicular neoplasm), Category V (suspicious for malignancy), Category VI (Malignant). If Cytology results shows Bethesda V or VI, then histology (categorical) will be performed.
Clinical outcomes: pathology at surgery (if surgery performed), | 6 months after randomization.
  Histologic examination (Categorical) will be performed to make diagnosis. Histology is a medical practice to review tissues under microscope to identify potential changes in a suspected tissue. The histological exam will help to diagnose if cancer is present or not and to find out the histologic type of the suspected tissue. The histologic types for thyroid cancer are as follows: Papillary, follicular, oncocytic, medullary, and anaplastic.
Clinical outcomes; Nodule size | Baseline and 6 months after randomization.
  If patient is on active monitoring, then the nodule size will be followed with ultrasound exams.
Score on selected domains of the ThyPRO short form instrument | 3 and 6 months post randomization
  The ThyPRO survey is a quality-of-life measure designed to evaluate how thyroid disease has affected the participant's life. Domains being used from this measure for the pilot study include symptoms (8 items), tiredness (2 items), and memory and concentration (3 items). Answer choices range from 1 (not at all) to 5 (very much) with higher scores indicating worse quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Louise Davies, MD, MS, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No